CLINICAL TRIAL: NCT04666402
Title: Integrated Diagnostics for Early Diagnosis of Liver Disease
Acronym: ID LIVER
Status: Recruiting | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Manchester (Other); University of Nottingham (Other); Innovate UK (Other Government)
Responsible Party: Sponsor
Other Study IDs: B00907
Record Dates: First submitted 2020-10-21; First posted 2020-12-14 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non-alcoholic Steatohepatitis; Alcoholic Liver Disease; Liver Fibroses
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases, Alcoholic; Liver Cirrhosis | interventions — Hematologic Tests; Polymorphism, Single Nucleotide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum for specific single nucleotide polymorphisms will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood tests for Single Nucleotide Polymorphisms — This extra test would be performed on participants assessed in the specialist liver clinic. This test would require an extra 5ml of blood to be taken at the time of routine blood tests for clinical purposes.
Diagnostic Test: Faecal microbiome analysis — This test will be undertaken for all participants who give consent and are assessed through the new liver care pathway, in the community liver assessment clinic. All participants will be given the equipment to take a stool sample at the time of presentation at the community liver assessment clinic and asked to return the sample to the clinic. The sample will be processed to remove genetic material so the microbiome can be identified.
Diagnostic Test: Serum for diagnostic biomarkers — Blood samples will be taken alongside blood taken for clinical assessment. In total, an extra 5ml of blood. These samples will be used to explore novel blood biomarkers using ELISA and mass-spectroscopy techniques in the University of Manchester.

SUMMARY:
This is an observational study that will explore the hypothesis that by combining data from patients with liver disease with novel blood biomarkers, single nucleotide polymorphism (SNP) analysis and faecal microbiome analysis. The Investigators will improve diagnosis of liver fibrosis compared to the current available diagnostic tools.

DETAILED DESCRIPTION:
Liver disease is a silent epidemic. Four in ten people in the North West are likely to have evidence of liver disease. A small but significant proportion of these patients develop scarring, leading to end-stage cirrhosis. All too frequently this is detected in very advanced stages, where treatment cannot reverse the condition. It is one of the UK's largest health challenges. At present clinicians use a wide range of single tests that individually struggle to identify disease and high-risk patients early.

The Investigators are implementing a new pathway for the assessment of patients with abnormal liver blood tests or high risk for liver disease. This novel pathway will allow assessment of patients in Community Liver Assessment Clinics (CLAC) with the expectation that only 20% of patients assessed would need to be seen in secondary care for further assessment. The investigators expect, to be assessing, 750 patients per year in this pathway. This pathway will bring together a large group of patients with liver disease. As part of the clinical assessment the investigators will be undertaking investigations to diagnose disease and assess extent. This will generate significant information, that the investigators currently use in isolation to make the aforementioned assessments. In this study, the investigators would like to bring together all this data into a curated database. To this end, the investigators would offer all patients who attend the CLAC for clinical need to enrol into the study. This would generate a database to combine all data, alongside some other, non-invasive tests, done alongside routine clinical tests.

This project will address this lack of answers by teaming up with innovative companies to make software that joins together a wide range of different tests to make an algorithm to detect disease earlier.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to Community Liver Assessment Clinic.
* Male or female > 18 years of age.
* Females will be non-pregnant and non-lactating.

Exclusion Criteria:

* Age < 18 years.
* Pregnancy/breast-feeding. Women of childbearing potential (not >2 years post- menopausal and/or not surgically sterilised) must have a negative blood serum pregnancy test.
* Isolated bilirubinaemia.
* Known pre-existing liver disease.
* Acutely unwell.
* Suspected malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending Community Liver Assessment Clinic within Manchester with deranged liver function tests, fatty liver on ultrasound or a history of alcohol excess
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in patient numbers requiring secondary care appointments for the investigation of advanced liver fibrosis. | At study completion; within 3 years
  Our project aims to identify patients with liver fibrosis in the community and only those with evidence of advanced fibrosis or cirrhosis being triaged on into secondary care hepatology services.

SECONDARY OUTCOMES:
To define the metrics involved in the diagnosis of advanced liver fibrosis or cirrhosis | At study completion; Within 3 years
  Through combining the data from basic clinical bloods such as LFTs, non-invasive scoring systems such as FIB-4 and NAFLD fibrosis scores along with the novel biomarkers, we will use this data through AI to develop algorithms that will aid the diagnosis of advanced fibrosis/cirrhosis.

CONTACTS AND LOCATIONS:
Overall Officials: Varinder Athwal, Principal Investigator — Manchester University NHS Foundation Trust/Manchester University
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No